CLINICAL TRIAL: NCT05243823
Title: Vaginal Estradiol Tablets (Vagifem®) and Endometrial Cancer Risk in the Treatment of Postmenopausal Vaginal Atrophy: A Register-based Cohort Study in Postmenopausal Women
Brief Title: Vaginal Estradiol Tablets (Vagifem®) and Endometrial Cancer Risk in the Treatment of Postmenopausal Vaginal Atrophy
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: VAG-4602; U1111-1270-0966 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-01-14; First posted 2022-02-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Danish cohort: Danish cohort starts on 1 January 2000 and ends on 31 December 2019. It consists of new users of low dose vaginal estrogens (LDVE) (split into Vagifem® and other LDVE products) in the study period, and a comparator group consisting of women using no hormone replacement therapy.
  Interventions: Drug: Vagifem®; Drug: Non-Vagifem® LDVE, Estradiol
- US cohort: US cohort starts on 1 January 2007 and ends on 31 December 2019. It consists of new users of low dose vaginal estrogens (LDVE) (split into Vagifem® and other LDVE products) in the study period, and a comparator group consisting of women using no hormone replacement therapy.
  Interventions: Drug: Vagifem®; Drug: Non-Vagifem® LDVE, Estradiol

INTERVENTIONS:
Drug: Vagifem® — According to local clinical practice - independent of inclusion in this study
Drug: Non-Vagifem® LDVE, Estradiol — According to local clinical practice - independent of inclusion in this study

SUMMARY:
The study will include data from a nationwide Danish cohort of postmenopausal women and the United States of America (US) cohort of postmenopausal women. The Danish nationwide cohort will be established through linkage of Danish national patient registries. The US cohort will be established based on data from US claims database, Truven. The aim of this study is to evaluate whether exposure to Vagifem® increases the rate of endometrial cancer in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 50-75 years at entry

Exclusion Criteria:

1. Endometrial cancer prior to entry
2. Any use of vaginal estrogen products prior to entry
3. Hysterectomy prior to entry

Ages: 50 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study population includes postmenopausal women split into two separate cohort studies from two countries - Denmark and US. The study population for both the Danish and the US cohort consists of new users of LDVE (split into Vagifem® and other LDVE products) in the study period, and a comparator group consisting of women using no hormone replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
First time occurrence of endometrial cancer (yes/no) during time in cohort from entry (start of treatment) to exit (end of study period, occurrence of any other cancer (except non-melanoma skin cancer), date of emigration or date of death) | From entry (day 0) to exit (upto 19 years)
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Soeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com